CLINICAL TRIAL: NCT00994461
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase 4 Study To Compare The Effect Of Celecoxib 100 Mg BID, Loxoprofen 60 Mg TID And Placebo On The Gastroduodenal Mucosa In Healthy Subjects
Brief Title: Study Of Celecoxib In Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3191345
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: Endoscopy
MeSH Terms: interventions — Celecoxib; loxoprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Celecoxib (Experimental)
  Interventions: Drug: Celecoxib
- Loxoprofen (Active Comparator)
  Interventions: Drug: Loxoprofen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 100mg tablet twice a day with meal for 2 weeks
  Arms: Celecoxib
Drug: Loxoprofen — Loxoprofen 60mg tablet three times a day with meal for 2 weeks
  Arms: Loxoprofen
Drug: Placebo — Placebo tablet three times a day with meal for 2 weeks
  Arms: Placebo

SUMMARY:
A study to confirm the superiority of celecoxib 100 mg BID to loxoprofen 60 mg TID in the incidence of gastroduodenal endoscopic ulcers after 2 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers

Exclusion Criteria:

* Endoscopic evidence of ulceration, erosion or active bleeding etc. in the esophagus, stomach, pylorus and/or duodenum prior to treatment endoscopy
* A history of gastrointestinal ulcer
* Any use of celecoxib, nonsteroidal anti-inflammatory drugs (including aspirin), anti-ulcer medication, antacids, systemic steroids or antibiotics within four weeks prior to the first dose of study medication

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Japan (3):
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo

REFERENCES:
- [Derived] Sakamoto C, Kawai T, Nakamura S, Sugioka T, Tabira J. Comparison of gastroduodenal ulcer incidence in healthy Japanese subjects taking celecoxib or loxoprofen evaluated by endoscopy: a placebo-controlled, double-blind 2-week study. Aliment Pharmacol Ther. 2013 Feb;37(3):346-54. doi: 10.1111/apt.12174. Epub 2012 Dec 10. PMID 23216412
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191345&StudyName=Study%20Of%20Celecoxib%20In%20Healthy%20Subjects

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 3 centers in Japan.
Groups:
- Celecoxib: Celecoxib 100 mg tablet twice a day with meal for 2 weeks
- Loxoprofen: Loxoprofen 60 mg tablet three times a day with meal for 2 weeks
Period: Overall Study
Arm/Group | Celecoxib | Loxoprofen | Placebo
Started | 76 | 76 | 37 (One subject was randomized but did not receive study drug.)
Completed | 74 | 75 | 37
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Loxoprofen | Placebo | Total
Number analyzed (Participants) | 76 | 76 | 37 | 189
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (9.65) | 57.8 (9.38) | 59.1 (9.18) | 57.5 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 26 | 135
  Male | 22 | 21 | 11 | 54
Helicobacter pylori (H. pylori) status [Number; unit: Participants]
  Positive | 32 | 33 | 16 | 81
  Negative | 44 | 43 | 21 | 108

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Gastroduodenal Ulcers
Description: The percentage of subjects who had gastroduodenal endoscopic ulcers after 2 weeks treatment (The number of subjects who had gastroduodenal endoscopic ulcers after 2 weeks treatment divided by participants multiplied by 100.) An ulcer is defined as any break in the mucosa at least 3 mm in diameter with unequivocal depth.
Time Frame: 2 weeks
Population: The modified-safety analysis set (m-SAF) consisted of all randomized subjects who received at least one dose of the study drug, and underwent endoscopy at baseline and at the end/discontinuation of treatment, as well.
Measure: Number; unit: Percent
Arm/Group | Celecoxib | Loxoprofen | Placebo
Number analyzed (Participants) | 74 | 76 | 37
Percent | 1.4 | 27.6 | 2.7
Statistical Analysis 1: Comparison: Celecoxib vs Loxoprofen; Hypothesis testing was conducted with significant p-value level of under 0.05; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) test stratified by H. pylori status was employed for the comparison of celecoxib and loxoprofen with placebo. The multiplicity of test was not adjusted because these comparisons were for the secondary objective; CMH test stratified by H. pylori status was employed. Continuous correction was used

2. Secondary Outcome: Incidence of Any Gastric, and Duodenal Ulcers
Description: The percentage of subjects who had gastric and duodenal endoscopic ulcers after 2 weeks treatment (The number of subjects who had gastric and duodenal endoscopic ulcers after 2 weeks treatment divided by participants multiplied by 100.) An ulcer is defined as any break in the mucosa at least 3 mm in diameter with unequivocal depth.
Time Frame: 2 weeks
Population: The m-SAF consisted of all randomized subjects who received at least one dose of the study drug, and underwent endoscopy at baseline and at the end/discontinuation of treatment, as well.
Measure: Number; unit: Percent
Arm/Group | Celecoxib | Loxoprofen | Placebo
Number analyzed (Participants) | 74 | 76 | 37
Percent
  Gastric ulcers | 0 | 25.0 | 2.7
  Duodenal ulcers | 1.4 | 5.3 | 0

3. Secondary Outcome: Incidence of Any Gastroduodenal, Gastric, and Duodenal Ulcers and/or Erosions
Description: The percentage of subjects who had gastroduodenal, gastric, and duodenal endoscopic ulcers and/or erosions after 2 weeks treatment (The number of subjects who had gastroduodenal, gastric, and duodenal endoscopic ulcers and/or erosions after 2 weeks treatment divided by participants multiplied by 100.) An ulcer is defined as any break in the mucosa at least 3 mm in diameter with unequivocal depth. An erosion is defined as a lesion producing a definite break in the mucosa with equivocal depth.
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Number; unit: Percent
Arm/Group | Celecoxib | Loxoprofen | Placebo
Number analyzed (Participants) | 74 | 76 | 37
Percent
  Gastroduodenal ulcers and/or erosions | 36.5 | 53.9 | 24.3
  Gastric ulcers and/or erosions | 35.1 | 53.9 | 24.3
  Duodenal ulcers and/or erosions | 4.1 | 5.3 | 0

4. Secondary Outcome: Post-treatment Gastroduodenal Endoscopic Scores (According to Mucosal Grading Scale)
Description: Number of subjects for each gastroduodenal endoscopic score (according to Mucosal Grading Scale) after 2 weeks treatment (Score 0 = normal mucosa (no visible lesions); Score 1 = 1 to 10 petechiae; Score 2 = more than 10 petechiae; Score 3 = 1 to 5 erosions; Score 4 = 6 to 10 erosions; Score 5 = 11 to 25 erosions; Score 6 = more than 25 erosions; Score 7 = ulcer)
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Celecoxib | Loxoprofen | Placebo
Number analyzed (Participants) | 74 | 76 | 37
Participants
  Score 0 | 38 | 33 | 22
  Score 1 | 8 | 2 | 6
  Score 2 | 1 | 0 | 0
  Score 3 | 22 | 19 | 8
  Score 4 | 4 | 1 | 0
  Score 5 | 0 | 0 | 0
  Score 6 | 0 | 0 | 0
  Score 7 | 1 | 21 | 1

5. Secondary Outcome: Number of Gastroduodenal Ulcers in Each Subject
Description: Number of subjects for each number of gastroduodenal endoscopic ulcers after 2 weeks treatment (An ulcer is defined as any break in the mucosa at least 3 mm in diameter with unequivocal depth.)
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Celecoxib | Loxoprofen | Placebo
Number analyzed (Participants) | 74 | 76 | 37
Participants
  0 ulcer | 73 | 55 | 36
  1 ulcer | 1 | 10 | 1
  2 ulcers | 0 | 5 | 0
  3 ulcers | 0 | 2 | 0
  4 ulcers | 0 | 0 | 0
  5 ulcers | 0 | 0 | 0
  6 ulcers | 0 | 1 | 0
  7 ulcers | 0 | 2 | 0
  8 ulcers | 0 | 1 | 0
  9 ulcers | 0 | 0 | 0
  10 or more ulcers | 0 | 0 | 0

6. Secondary Outcome: Number of Gastroduodenal Erosions in Each Subject
Description: Number of subjects for each number of gastroduodenal endoscopic erosions after 2 weeks treatment (An erosion is defined as a lesion producing a definite break in the mucosa with equivocal depth.)
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Celecoxib | Loxoprofen | Placebo
Number analyzed (Participants) | 74 | 76 | 37
Participants
  0 erosion | 47 | 41 | 29
  1 erosion | 14 | 13 | 5
  2 erosions | 4 | 3 | 1
  3 erosions | 5 | 9 | 2
  4 erosions | 0 | 4 | 0
  5 erosions | 0 | 3 | 0
  6 erosions | 2 | 1 | 0
  7 erosions | 1 | 1 | 0
  8 erosions | 0 | 1 | 0
  9 erosions | 0 | 0 | 0
  10 or more erosions | 1 | 0 | 0

7. Secondary Outcome: Incidence of Treatment-emergent, All-causality GI Body System Adverse Events
Description: The percentage of subjects who had treatment-emergent, all-causality gastrointestinal body system adverse events after 2 weeks treatment (The number of subjects who had treatment-emergent, all-causality gastrointestinal body system adverse events after 2 weeks treatment divided by participants multiplied by 100.)
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Number; unit: Percent
Arm/Group | Celecoxib | Loxoprofen | Placebo
Number analyzed (Participants) | 74 | 76 | 37
Percent | 24.3 | 47.4 | 16.2

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Celecoxib | Loxoprofen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76 | 0/37
Other Adverse Events (participants affected / at risk) | 19/76 | 37/76 | 8/37
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=76) | Loxoprofen (N=76) | Placebo (N=37)
Abdominal discomfort (Gastrointestinal disorders) | 2 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 2 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 5 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 4 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 8 | 28 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.